CLINICAL TRIAL: NCT01844843
Title: Evaluation With OFDI of Strut Coverage of Terumo New Drug Eluting Stent (Development Code TCD-10023) With Biodegradable Polymer at 1, 2 and 3 Months
Brief Title: Optical Frequency Domain Imaging (OFDI) Assessed Strut Coverage of New Terumo DES
Acronym: DISCOVERY123
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T121E4
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease
Keywords: Drug eluting stents; coronary artery disease; Percutaneous Coronary Intervention; Tomography, Optical Coherence
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TCD-10023 drug eluting stent (Experimental): All patients will be treated with the new Drug eluting stent TCD-10023
  Interventions: Device: TCD-10023 drug eluting stent

INTERVENTIONS:
Device: TCD-10023 drug eluting stent — Implantation of new drug eluting stent in coronary artery lesions

SUMMARY:
Purpose of this study is to evaluate, after implantation of a drug eluting stent (DES), coverage of the stent struts by new tissue. The evaluation will be performed by means of intravascular imaging technology (optical frequency domain imaging, OFDI). Renewed tissue coverage over the implanted stent struts prevents direct contact between blood and metal/polymer, which could lead to adverse events: patients need to take blood-thinning drugs to prevent these events. Ous new stent has drug and polymer only on the outside of the stent, and the polymer is degraded by the body leaving a bare metal stent after 3-4 months. This should allow fast coverage of the struts, and might allow to reduce duration of the supportive medical treatment. Our hypothesis is that <20% of the struts remain uncovered at 3 months after implantation, as assessed by OFDI.

DETAILED DESCRIPTION:
We will enroll patients with multiple coronary lesions, which, as is routine practice, will be treated with the new DES in 2 sessions (second one approximately 3-5 weeks after the first one). We will assess lesions by OFDI after the implantation and at the time of 3 months follow-up, when we will ask patients to undergo a coronary angiography. Patients will then have a follow-up contact at 1 year after initial implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Patients is a suitable candidate for Percutaneous Coronary Intervention (PCI)
* Patient has multi-vessel disease with ≥2 de-novo lesions in native coronary arteries suitable for treatment with TCD-10023 DES
* Target lesions are suitable for OFDI examination;
* Patient requires staged procedure between 3-5 weeks after baseline procedure, according to investigator's judgement
* Target vessel reference diameter is between 2.5 - 4.0 mm (visual assessment)
* Patient has provided written informed consent
* Patient is affiliated to social security or equivalent system (France only)

Exclusion Criteria:

* - Patient has known allergy to sirolimus, cobalt, chromium, nickel, or contrast agent (that cannot be adequately premedicated)
* Patient is not a suitable candidate for use of Dual Anti-Platelet Therapy (DAPT) because of active or recent bleedings or for use of vitamin K antagonist, like warfarin, dabigatran, rivaroxaban or acenocoumarol;
* Patient is presenting with ST-segment elevated MI (STEMI) at baseline procedure
* Patient has Killip-class > 1 at admission
* Patient is in cardiogenic shock
* Patient is a female of childbearing potential
* Patient has life expectancy of less then 1 year
* Patient is expected to undergo major surgery within 3 months
* Patient has Left Main disease ≥ 50%
* Target lesion at bifurcation requiring 2 stents technique
* Target lesions are severely calcified
* Target lesion is located within 3 mm of aorta-ostium
* Patient has renal failure defined as estimated Glomerular Filtration Rate (eGFR) <50 mL/min/1.73m²
* Target lesions require preparation other than balloon pre-dilatation
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints; Note: Trials requiring extended follow-up for products that were investigational, but have become commercially available since then, are not considered investigational trials
* In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study
* Patient is under judicial protection (France only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
OFDI assessed percent stent strut coverage | 3 months post procedure.

SECONDARY OUTCOMES:
% stent strut coverage | at 1 and 2 months
% stented lesions with >10% uncovered struts | at 1, 2, 3 months
% of stented lesions with >20% uncovered stent struts | at 1, 2, 3 months
% of acquired mal-apposed stent struts | at 1, 2, 3 months
amount (mm³) of in-stent intimal hyperplasia | at 1, 2, 3 months
amount (mm³)of in-segment hyperplasia | at 1, 2, 3 months
neo-intimal thickness (µm) | at 1, 2, 3 months
in-stent late lumen loss (mm) assessed by Quantitative Coronary Angiography (QCA) | at 3 months
In-segment late lumen loss (mm) assessed by QCA | at 3 months
Target Lesion revascularization (TLR) | at 1, 3, 12 months
Target Lesion Failure (TLF - composite of cardiac death, Myocardial infarction, TLR | at 1, 3, 12 months
Target Vessel Revascularization (TVR) | at 1, 3, 12 months
Major Cardiac Adverse Events (MACE) defined as cardiac death, Q wave and non-Q wave Myocardial Infarction (MI) , emergent coronary artery bypass surgery, or target vessel revascularization (TVR) | at 1, 3, 12 months
Stent thrombosis | at 1, 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Smits, MD, Study Chair — Maasstad hospital, Rotterdam, the Netherlands; Bernard Chevalier, MD, Study Chair — Cardiovascular Institute Paris Sud, Massy, France
Locations (6):
- France (2):
  - Cardiovascular Institute Paris Sud (ICPS), Massy
  - CHU Rangueil, Toulouse
- LMU, München, Germany
- Netherlands (3):
  - MCL, Leeuwarden
  - Erasmus, Rotterdam
  - Maasstadziekenhuis, Rotterdam

REFERENCES:
- [Derived] Chevalier B, Smits PC, Carrie D, Mehilli J, Van Boven AJ, Regar E, Sawaya FJ, Chamie D, Kraaijeveld AO, Hovasse T, Vlachojannis GJ. Serial Assessment of Strut Coverage of Biodegradable Polymer Drug-Eluting Stent at 1, 2, and 3 Months After Stent Implantation by Optical Frequency Domain Imaging: The DISCOVERY 1TO3 Study (Evaluation With OFDI of Strut Coverage of Terumo New Drug Eluting Stent With Biodegradable Polymer at 1, 2, and 3 Months). Circ Cardiovasc Interv. 2017 Dec;10(12):e004801. doi: 10.1161/CIRCINTERVENTIONS.116.004801. PMID 29246909